CLINICAL TRIAL: NCT00035425
Title: A Randomized, Double-Blind Trial Comparing Linezolid To Vancomycin In The Empiric Treatment Of Febrile Neutropenic Oncology Patients With Suspected Gram-Positive Infections
Brief Title: Treatment of Neutropenic Patients With Fever Who Are Suspected to Have A Gram Positive Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: M12600079; A5951059
Record Dates: First submitted 2002-05-03; First posted 2002-05-06 (Estimated); Last update posted 2009-12-01 (Estimated); Status verified 2009-11

CONDITIONS: Febrile Neutropenia
MeSH Terms: conditions — Febrile Neutropenia | interventions — Linezolid; Vancomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A. (Experimental): Patients will be stratified according to the use of prophylactic antibiotics. Both groups may receive open-label gram-negative coverage with either ceftazidime, aztreonam, and/or aminoglycosides (gentamicin, tobramycin, amikacin). Subjects will receive study medication intravenously every 12 hours for 7 to 28 days.
  Interventions: Drug: linezolid
- B. (Experimental)
  Interventions: Drug: vancomycin

INTERVENTIONS:
Drug: linezolid — 600mg every 12 hours
  Other Names: Zyvox
  Arms: A.
Drug: vancomycin — 1gm every 12 hours. The dose of vancomycin intravenously may be adjusted for renal function, but the patient must be able to receive a 300 mL volume of intravenous fluid at the assigned dosing times of every 12 hours.
  Arms: B.

SUMMARY:
This study will treat patients who have fever and neutropenia (after cancer chemotherapy) that is possibly due to a specific bacteria (gram positive bacteria).

ELIGIBILITY:
Inclusion Criteria:

Patients must have neutropenia (ANC less than 500) with fever (oral temp 38.3 C).

Patients must have a cancer with recent chemotherapy and risks factors for gram positive infections.

Exclusion Criteria:

Patients with fever due to known causes. Patients with HIV. Patients with recent bone marrow transplant. Patients with an infected indwelling catheter that cannot be removed. Patients who have received more than one day of another antibiotic before entering the trial.

Patients with endocarditis, osteomyelitis, meningitis, CNS infections.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2001-11; Study Completion 2002-11 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy of linezolid when administered intravenously as compared to intravenously administered vancomycin in the empiric treatment of oncology patients with febrile neutropenia with suspected gram-positive infections. | 7-28 days

SECONDARY OUTCOMES:
Microbiologic outcome | 7-28 days
Pathogen eradication (eradication rates of individual pathogens) | 7-28 days
Defervescence (defined as Tmax orally or rectally) | 7-28 days
Time to defervescence | 7-28 days
Resolution of neutropenia (return of ANC to >500 cells/mm3) | 7-28 days
Time to resolution of neutropenia | 7-28 days
Mortality rate (survival at 7 days after the end of therapy) | 7-28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (8):
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Springfield, Illinois
  - Pfizer Investigational Site, The Bronx, New York
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Federal Way, Washington
  - Pfizer Investigational Site, Lakewood, Washington
  - Pfizer Investigational Site, Tacoma, Washington
- Argentina (3):
  - Pfizer Investigational Site, Buenos Aires
  - Pfizer Investigational Site, Córdoba
  - Pfizer Investigational Site, Mendoza
- Brazil (2):
  - Pfizer Investigational Site, Porto Alegre, Rio Grande do Sul
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Santiago, Chile
- Colombia (2):
  - Pfizer Investigational Site, Bogotá, Bogota. DC
  - Pfizer Investigational Site, Medellín
- Pfizer Investigational Site, Helsinki, Finland
- Mexico (3):
  - Pfizer Investigational Site, Zapopan, Jalisco
  - Pfizer Investigational Site, Monterrey, Nuevo León
  - Pfizer Investigational Site, Mexico City
- Pakistan (2):
  - Pfizer Investigational Site, Lahore, Punjab Province
  - Pfizer Investigational Site, Karachi
- Pfizer Investigational Site, Lima, Lima Province, Peru
- Venezuela (2):
  - Pfizer Investigational Site, Caracas, Distrito Federal
  - Pfizer Investigational Site, Caracas
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=M12600079&StudyName=Treatment%20of%20Neutropenic%20Patients%20With%20Fever%20Who%20Are%20Suspected%20to%20Have%20A%20Gram%20Positive%20Infection%20